CLINICAL TRIAL: NCT07337408
Title: Characterization of Weaning Practices in ICUs of Global South Countries: A Prospective Observational Study
Brief Title: Characterization of Weaning Practices in ICUs of Global South Countries
Status: Not yet recruiting | Type: Observational
Sponsor: Hospital do Coracao (Other)
Responsible Party: Sponsor
Other Study IDs: GS Wean - Observational
Record Dates: First submitted 2025-12-23; First posted 2026-01-13 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2026-02

CONDITIONS: Weaning From Mechanical Ventilation; Weaning Failure; Weaning From Mechanical Ventilation, Extubation
Keywords: Weaning from mechanical ventilation; Weaning Failure; Weaning from mechanical ventilation, extubation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective observational study to be conducted in intensive care units of Global South countries. Patients on mechanical ventilation for more than 12 hours who have initiated the weaning process and for whom the attending team plans extubation within the next 6 hours will be included. Data will be collected for each patient during the first 7 days after extubation, with follow-up until hospital discharge or death. We plan to conduct the study in intensive care units from Global South countries (low- and middle-income countries predominantly located in the Southern Hemisphere, though some in the Northern Hemisphere are also considered).

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years.
* Receiving care at an intensive care unit.
* Endotracheal intubation.
* Mechanical ventilation for 12 hours or more.
* First separation attempt, as defined in the WIND Classification - "Separation attempt from mechanical ventilation: an spontaneous breathing trial with or without extubation, or an extubation directly performed without identified spontaneous breathing trial (whatever the type: planned or unplanned extubation)" - planned to occur in the next 6 hours or that occurred less than 2 hours ago.

Exclusion Criteria:

* Patients with prior extubation failure.
* Patients with prior spontaneous breathing trial failure.
* Patients unable to obey commands.
* Neuromuscular disease or cervical spinal cord injury.
* Tracheostomy.
* Do-not-resuscitate order or contraindication for reintubation.
* Lack of informed consent.
* Terminal extubation.
* Previously included in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients receiving mechanical ventilation for more than 12 hours who are planning to undergo the first separation attempt from the invasive mechanical ventilation (as defined in the WIND Classification) in the next 6 hours or that has undergone a separation attempt less than 2 hours ago will be included.
Sampling Method: Non-Probability Sample
Enrollment: 900 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2027-03 (Estimated); Study Completion 2027-04 (Estimated)

PRIMARY OUTCOMES:
Extubation failure within 7 days. | 7 days.
  Defined as reintubation or death within 7 days after extubation.

SECONDARY OUTCOMES:
Extubation within 28 days. | 28 days.
  Defined as extubation within 28 days after first separation attempt.
Intensive care unit length of stay. | At intensive care unit discharge, up to 28 days.
  Defined as the number of days from the time of first separation attempt until discharge from the intensive care unit.
Hospital length of stay. | At hospital discharge, up to 28 days.
  Defined as the number of days from the time of first separation attempt until discharge from the hospital.
Reintubation or death within 28 days. | 28 days.
  Defined as composite criterion of reintubation or death within 28 days after first separation attempt.
Intensive care unit mortality. | At intensive care unit discharge, up to 28 days.
  Defined as mortality from the time of first separation attempt until discharge from the intensive care unit.
Hospital mortality. | At hospital discharge, up to 28 days.
  Defined as mortality from the time of first separation attempt until discharge from the hospital.
Number of spontaneous breathing trials. | 28 days.
  Defined as the number of spontaneous breathing trials performed after first separation attempt.
WIND classification. | 28 days.
  Group 1 (short weaning): the first separation attempt resulted in a termination of the weaning process within 24 hours (successful separation or early death). • Group 2 (difficult weaning): weaning was terminated after more than 1 day but in less than 1 week after the first separation attempt (successful separation or death). • Group 3 (prolonged weaning): weaning was still not terminated 7 days after the first separation attempt (by success or death).